CLINICAL TRIAL: NCT00247533
Title: The Early Diagnosis and Prevention of Ischemic Stroke and Cognition Decline Associated With Coronary Artery Disease Combined With Cerebral Artery Stenosis or Arrhythmia by 24-Hour Simultaneous Recorder of Electrocardiograph and Electroencephalography
Brief Title: Cerebral Artery Stenosis, Coronary Artery Disease and Arrhythmia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: FEMH-E-940004
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2005-08

CONDITIONS: Stroke; Coronary Artery Disease; Arrhythmia
Keywords: coronary disease; cerebrovascular disorders; angiography; cerebral ischemia; intracranial atherosclerosis; Coronary artery disease; cerebral artery stenosis; percutaneous coronary balloon angioplasty; coronary artery bypass surgery; ischemic stroke; electrocardiograph; electroencephalograph; Nuclear brain scan; cognition decline; atrial fibrillation; undetermined ischemic stroke
MeSH Terms: conditions — Stroke; Coronary Artery Disease; Arrhythmias, Cardiac; Coronary Disease; Cerebrovascular Disorders; Brain Ischemia; Intracranial Arteriosclerosis; Ischemic Stroke; Atrial Fibrillation

INTERVENTIONS:
Procedure: Digital subtraction angiography and 24-hour simultaneous recorder of electrocardiograph

SUMMARY:
There are many reports about the association of coronary artery disease (CAD) and cerebral artery stenosis (CAS), which had been proved to induce stroke and cognition decline after the revascularization including coronary bypass surgery (CABG) or percutaneous coronary intervention. Perfusion defect on nuclear brain scan is also noted to correlate with these neurological complications. On the other hand, the perioperative arrhythmia and following cerebral embolism was also attributed to be one factor inducing such neurological hazards.

In the patients with coexistent CAD and CAS (1st group), and also the patients scheduled for CABG or percutaneous coronary intervention (PCI) (2nd group), we, the researchers at Far Eastern Memorial Hospital, attempted to integrate all the parameters mention above, including angiography of coronary and cerebral system, quantitative analysis of nuclear brain scan, biochemical profile, and signals of a new ambulatory device which could record the electrocardiograph (ECG) and electroencephalograph (EEG) simultaneously, in order to define the correlation between them. A chorological relation between EEG signals and ECG signals is our first target to be worked out. Thereafter, we hope to establish a regression model of all involved parameters according to the relation. Such a model, we believe, is essential not only to explain the post-CABG neurological complications, but to prevent them.

Furthermore, for the undetermined ischemic stroke patients who had no obvious culprit artery or embolism source, the paroxysmal arrhythmia had long been regarded as the cause. Whether a paroxysmal atrial fibrillation, which had not been disclosed by routine ECG, could induce most of such a stroke is still not known. With this new ambulatory device which could record the electrocardiograph (ECG) and electroencephalograph (EEG) simultaneously, we want to answer the question.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery stenosis >50% and either carotid or brain artery stenosis > 50%

Exclusion Criteria:

* Creatinine > 2.0 mg/dL
* Co-morbidity
* ER
* A letter of authorization is not given

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: A H Li, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taipei, Taiwan